CLINICAL TRIAL: NCT05553938
Title: Renal Mechanistic Effects of Acute and Chronic Empagliflozin in Heart Failure
Brief Title: Effects of Acute and Chronic Empagliflozin Heart Failure
Acronym: EMPA HF
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2000033412
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Double blind placebo controlled, with crossover for placebo patients to active drug at 6 weeks. (At 6 weeks, participants are unblinded, and participants who received placebo will receive study drug.)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin (Experimental): Empagliflozin 10 mg daily for weeks 1-6
  Interventions: Drug: Empagliflozin 10 mg
- Placebo, Then Empagliflozin (Experimental): Participants first receive matching placebo daily for weeks 1-6, then will receive Empagliflozin 10 mg daily for weeks 7-12
  Interventions: Drug: Empagliflozin 10 mg; Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin 10 mg — Empagliflozin 10mg
Drug: Placebo — Empagliflozin matched placebo tablet
  Arms: Placebo, Then Empagliflozin

SUMMARY:
This is a 60-patient randomized, double-blind, placebo-controlled mechanistic study to understand the utility of empagliflozin in worsening heart failure (HF) patients with or without diabetes. Participants will be randomized to empagliflozin or placebo for 6 weeks, followed by a crossover of placebo patients to active therapy at 6 weeks-12 weeks.

DETAILED DESCRIPTION:
This is a 60-patient randomized, double-blind, placebo-controlled mechanistic study to understand the utility of empagliflozin in worsening heart failure (HF) patients with or without diabetes.

The broad study design aims to evaluate change in gold standard determined body fluid spaces, sodium avidity, and cardio-renal biomarkers longitudinally in patients treated with placebo vs. empagliflozin over a 6 week period. Primary analysis of the randomized intervention will occur during the 6 week double blind period. Crossover of placebo patients to active therapy from 6-12 weeks will provide additional exploratory mechanistic data at low incremental cost and provide added benefit to enrollment of the study.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of worsening heart failure (worsening of congestive symptoms with current therapies) in the opinion of the investigator.
* A planned outpatient diuretic intervention (either up-titration of loop or addition of thiazide diuretic) for worsening heart failure per treating clinician. Diuretic intervention can occur via an unplanned in person visit (e.g., outpatient ambulatory clinic, emergency department, same day access visit) or via a telephone encounter (e.g., patient calling the clinic with reported weight gain and SOB that is prescribed uptitration of diuretic therapy).
* Estimated or reported weight gain of at least 5 lbs.
* Chronic daily oral loop diuretic dose ≥ 20mg furosemide equivalents for at least one month prior to enrollment
* Estimated GFR (eGFR) ≥ 20 mL/min/1.73 m2
* Age ≥ 18 years old
* Signed informed consent
* English speaking participants only

Exclusion Criteria:

* Need for heart failure hospitalization at the time of randomization
* Current use or plan to initiate renal replacement therapy
* Significant bladder dysfunction or urinary incontinence
* Inability to comply with the serial urine collection procedures
* Chronic use of natriuretic doses of thiazide diuretics (≥50mg hydrochlorothiazide or equivalent)
* Critical stenotic valvular disease, complex congenital heart disease or prior heart transplant
* History of type 1 diabetes, diabetic ketoacidosis, "brittle" diabetes or frequent hypoglycemia or severe hypoglycemic episodes requiring emergent intervention (ER visit or EMS response, glucagon administration or forced oral carbs) in the last 6 months
* History of or current urosepsis or frequent urinary tract infections
* Anemia with hemoglobin <8g/dL (due to required phlebotomy for the study) or active bleeding
* Pregnancy or breastfeeding
* Appears unlikely or unable to participate in the required study procedures, as assessed by the study PI, study coordinator, or designee (ex: clinically-significant psychiatric, addictive, or neurological disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-04 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Natriuretic effect of empagliflozin or placebo as an adjuvant to loop diuretic therapy | Day 1
  The natriuretic effect (urine sodium concentration) of each arm with loop diuretic therapy will be measured by the mmols of sodium excreted on day 1.
Change in plasma volume from baseline to 7 days | Day 1 and Day 7
  Chronic effects of empagliflozin or placebo to the loop diuretic will be assessed by measuring the change in plasma volume [ml] from Day 1 to Day 7, using I-131 albumin
Change in total body water from baseline to 7 days | Day 1 and Day 7
  Chronic effects of empagliflozin or placebo to the loop diuretic will be assessed by measuring the change in total body water [liters] from Day 1 to Day 7, using heavy water [D2O)

SECONDARY OUTCOMES:
Change in Chronic effects of empagliflozin vs placebo on plasma volume | Day 1 and day 42
  Chronic effects of empagliflozin vs placebo on change in plasma volume [ml] will be measured on Day 1 and Day 42, using I-131 albumin
Change in Chronic effects of empagliflozin vs placebo on change in total body water | Day 1 and day 42
  Chronic effects of empagliflozin vs placebo on change in total body water [liters] will be measured on Day 1 and Day 42, using heavy water [D2O]
Change in Chronic effects of empagliflozin on change in plasma volume during the open label extension. | Day 1 up to Day 84
  Changes in plasma volume[ml] from Day 1 to Day 84 will be assessed during the open label extension, using I-131 albumin
Change in Chronic effects of empagliflozin on change in total body water during the open label extension. | Day 1 up to Day 84
  Changes in total body water [liters] from Day 1 to Day 84 will be assessed during the open label extension, using heavy water [D2O]

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Testani, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No